CLINICAL TRIAL: NCT04720170
Title: Revascularization of the Lateral Plantar Artery and Anterior Pedal Loop of the Foot as Treatment for Diabetic Peripheral Neuropathy.
Brief Title: Exploratory Study of the Efficacy of Standard of Care Revascularization of the Lower Extremity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diabetes and Glandular Disease Clinic (Industry)
Collaborators: Modern Vascular, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBMK-001
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes; Type 1 Diabetes; Type 2 Diabetes; Neuropathy; Diabetic Peripheral Neuropathy; Peripheral Artery Disease; PAD
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: 26 week, single arm, single site
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): This is a 26 week, single arm, single-site, Investigator-initiated, exploratory trial evaluating the efficacy of the standard of care revascularization of the lower extremity with the addition of revascularization of the lateral plantar artery and anterior pedal loop of the foot as treatment for participants with PAD, diabetic neuropathy and have a clinical diagnosis of type 1 or type 2 diabetes whose main symptoms are numbness and/or tingling of the feet with or without pain.
  Interventions: Procedure: Revascularization

INTERVENTIONS:
Procedure: Revascularization — Angiogram and IVUS with revascularization of the lateral plantar artery and pedal arch on target foot.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the standard of care revascularization of the lower extremity with the addition of revascularization of the lateral plantar artery and anterior pedal loop of the foot as treatment for diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
This is a 26 week, single arm, single-site, Investigator-initiated, exploratory trial evaluating the efficacy of the standard of care revascularization of the lower extremity with the addition of revascularization of the lateral plantar artery and anterior pedal loop of the foot as treatment for participants with PAD, diabetic neuropathy and have a clinical diagnosis of type 1 or type 2 diabetes whose main symptoms are numbness and/or tingling of the feet with or without pain.

Participants who satisfy eligibility criteria may undergo standard of care revascularization of one lower extremity as required, with the addition of revascularization of the lateral plantar artery and anterior pedal loop followed by a 26-week follow-up phase. Standard of Care revascularization will be performed in any limb with ≥ 50% stenosis as determined by intra-vascular ultrasound (IVUS) at the time of planned study intervention.

Participants will be evaluated prior to intervention and at 2, 4, 14 and 26 weeks after the pedal loop intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 30 to 80 years (inclusive at first screening visit)
2. Clinical diagnosis of type 1 or type 2 diabetes as diagnosed by HbA1c ≥ 6.5% or current treatment
3. Clinical signs and symptoms of diabetic peripheral neuropathy bilaterally affecting the lower extremities, in the investigator's opinion, which may include neuropathic symptoms (e.g., numbness, tingling, burning sensation, sharp pains, sensitivity to touch) and decreased distal sensation (e.g., decreased vibration, pinprick or pain sensation, monofilament)
4. HbA1c ≤ 11% (historical results allowed if performed within the past 90 days)
5. Females of child-bearing potential who are willing to use contraceptive measures to prevent pregnancy for the duration of the study
6. Willing to attend all scheduled study visits and undergo all study procedures
7. Clinical diagnosis of Peripheral Artery Disease (PAD)
8. Be able to understand, speak, read and write English
9. Have medical insurance or financial means to cover the cost of the revascularization procedure and follow-up visits with the Interventional Radiologist

Exclusion Criteria:

1. Inability to undergo angiogram with revascularization
2. Unilateral neuropathic findings or symptoms
3. Vitamin B-12 level < 400 pg/ml (historical results allowed if performed within the past 30 days) *
4. Known causes of peripheral neuropathy other than diabetes, e.g., Amyloidosis, Tangier disease, Fabry's disease, hereditary sensory autonomic neuropathy, alcohol-related neuropathy, drug-induced neuropathy (e.g., chemotherapy, antibiotics, anti-retroviral agents, other neurotoxic agents) hypothyroidism that is not well controlled, rheumatoid arthritis or autoimmune disorders requiring treatment with corticosteroids, anti-tumor necrosis factor or immune-modulating medicines
5. Known history of Hepatitis B, C, or HIV
6. Lower limb amputation, including toe
7. Lower extremity inoperable occlusive vascular disease
8. Inability to provide informed consent
9. History of bleeding disorders
10. History of diabetic ulcers to the lower extremities
11. History of any surgical bypass of the lower extremities prior to randomization
12. History of previous revascularization of the lower extremities prior to randomization
13. End Stage Renal Disease (ESRD) requiring or on dialysis
14. Thyroid Stimulating Hormone -TSH >10.0 uu/mL*
15. Potassium > 5.5 mmol/L. *
16. Calcium < 8.5 mg/dL or > 11mg/dL *
17. Hemoglobin < 9.0 g/dL *
18. Female that is pregnant, breastfeeding or intends to become pregnant during the study period
19. Clinically significant abnormal ECG findings, in the opinion of the Investigator
20. Participation in another clinical trial with investigational drug or device at time of screening
21. Any other clinically significant disorders or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with the protocol requirements

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Intra-epidermal Nerve Fiber Density | 26 weeks
  Change from baseline in intra-epidermal nerve fiber density (IENFD) via skin biopsy of the revascularized foot over the extensor digitorum brevis muscle (EDBM) at week 26.

SECONDARY OUTCOMES:
Intra-epidermal Nerve Fiber Density | 14 and 26 weeks
  Number and percent of participants whose IENFD have increased by at least 20% from baseline
Utah Early Neuropathy Scale | 14 and 26 weeks
  Number and percentage of participants with improvement on Utah Neuropathy Scale (UENS)
Sural Nerve Action Potential Amplitude | 14 and 26 weeks
  Number and percentage of participants with improvement of sural nerve action potential amplitude
Sudoscan | 14 and 26 weeks
  Number and percentage of participants with 20% improvement on Sudoscan
Intra-epidermal Nerve Fiber Density | 14 weeks
  Number and percentage of participants with improvement of intra-epidermal nerve fiber density
Neuropathic Pain Syndrome Inventory | 14 and 26 weeks
  Improvement in quality of life as measured by the Neuropathic Pain Syndrome Inventory
Patency of Lateral Plantar Artery | 14 and 26 weeks
  Number and percentage of participants with patency of lateral plantar artery per ultrasound

OTHER OUTCOMES:
Medial Plantar Sural Nerve Action Potential Amplitude | 14 and 26 weeks
  Number of participants with 20% change in medial plantar sural nerve action potential amplitude (SNAP) via nerve conduction study

CONTACTS AND LOCATIONS:
Overall Officials: Dallas Broadway, MD, Principal Investigator — Modern Vascular, LLC; Mark S Kipnes, MD, Principal Investigator — Diabetes and Glandular Disease Clinic, P.A.
Locations (1):
- Diabetes and Glandular Disease Clinic, P.A., San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and Informed Consent
Supporting Information: Study Protocol, ICF
Time Frame: Starting 6 months after publication

REFERENCES:
- [Result] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Result] Cameron NE, Eaton SE, Cotter MA, Tesfaye S. Vascular factors and metabolic interactions in the pathogenesis of diabetic neuropathy. Diabetologia. 2001 Nov;44(11):1973-88. doi: 10.1007/s001250100001. PMID 11719828
- [Result] Ibrahim S, Harris ND, Radatz M, Selmi F, Rajbhandari S, Brady L, Jakubowski J, Ward JD. A new minimally invasive technique to show nerve ischaemia in diabetic neuropathy. Diabetologia. 1999 Jun;42(6):737-42. doi: 10.1007/s001250051222. PMID 10382594
- [Result] Malik RA, Masson EA, Sharma AK, Lye RH, Ah-See AK, Compton AM, Tomlinson DR, Hanley SP, Boulton AJ. Hypoxic neuropathy: relevance to human diabetic neuropathy. Diabetologia. 1990 May;33(5):311-8. doi: 10.1007/BF00403326. PMID 2376302
- [Result] Newrick PG, Wilson AJ, Jakubowski J, Boulton AJ, Ward JD. Sural nerve oxygen tension in diabetes. Br Med J (Clin Res Ed). 1986 Oct 25;293(6554):1053-4. doi: 10.1136/bmj.293.6554.1053. PMID 3094772
- [Result] Ram Z, Sadeh M, Walden R, Adar R. Vascular insufficiency quantitatively aggravates diabetic neuropathy. Arch Neurol. 1991 Dec;48(12):1239-42. doi: 10.1001/archneur.1991.00530240043016. PMID 1845025
- [Result] Singleton JR, Bixby B, Russell JW, Feldman EL, Peltier A, Goldstein J, Howard J, Smith AG. The Utah Early Neuropathy Scale: a sensitive clinical scale for early sensory predominant neuropathy. J Peripher Nerv Syst. 2008 Sep;13(3):218-27. doi: 10.1111/j.1529-8027.2008.00180.x. PMID 18844788
- [Result] Tesfaye S, Harris N, Jakubowski JJ, Mody C, Wilson RM, Rennie IG, Ward JD. Impaired blood flow and arterio-venous shunting in human diabetic neuropathy: a novel technique of nerve photography and fluorescein angiography. Diabetologia. 1993 Dec;36(12):1266-74. doi: 10.1007/BF00400804. PMID 8307254
- [Result] Veves A, Donaghue VM, Sarnow MR, Giurini JM, Campbell DR, LoGerfo FW. The impact of reversal of hypoxia by revascularization on the peripheral nerve function of diabetic patients. Diabetologia. 1996 Mar;39(3):344-8. doi: 10.1007/BF00418351. PMID 8721781
- [Result] Young MJ, Veves A, Walker MG, Boulton AJ. Correlations between nerve function and tissue oxygenation in diabetic patients: further clues to the aetiology of diabetic neuropathy? Diabetologia. 1992 Dec;35(12):1146-50. doi: 10.1007/BF00401368. PMID 1478366
- [Result] Young MJ, Veves A, Smith JV, Walker MG, Boulton AJ. Restoring lower limb blood flow improves conduction velocity in diabetic patients. Diabetologia. 1995 Sep;38(9):1051-4. doi: 10.1007/BF00402174. PMID 8591818
- See also: PubMed ID:11719828 — https://doi.org/10.1007/s001250100001
- See also: PubMed ID:10382594 — https://doi.org/10.1007/s001250051222
- See also: PubMed ID:2376302 — https://doi.org/10.1007/BF00403326
- See also: PubMed ID:3094772 — https://doi.org/10.1136/bmj.293.6554.1053
- See also: PubMed ID:8307254 — https://doi.org/10.1007/BF00400804
- See also: PubMed ID:8721781 — https://doi.org/10.1007/BF00418351
- See also: PubMed ID:1478366 — https://doi.org/10.1007/BF00401368
- See also: PubMed ID:8591818 — https://doi.org/10.1007/BF00402174